CLINICAL TRIAL: NCT02237638
Title: A Phase I Open-label Clinical Trial, Evaluating the Therapeutic Vaccine hVEGF26-104/RFASE in Patients With Advanced Solid Tumors
Brief Title: Phase I Study on VEGF Vaccination in Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Immunovo B.V. (Unknown)
Responsible Party: Principal Investigator, S. Derks, Medical Oncologist, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL45279.000.13
Record Dates: First submitted 2014-08-15; First posted 2014-09-11 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Cancer
Keywords: VEGF; Vaccine; Angiogenesis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hVEGF26-104/RFASE vaccination (Experimental): hVEGF26-104/RFASE is investigated in dose escalation in which hVEGF26-104 is escalated from 62.5 ug to 500 ug and RFASE is given in a fixed dose of 20 mg. Three patients are treated at each dose level. If 0 of the 3 patients are observed to have DLT, the dose level is escalated one step for the next cohort. If 1 of the 3 patients shows DLT, 3 additional patients are treated at that dose level. If none of these show DLT, the dose level is escalated for the next cohort; otherwise, the prior dose level is defined as the MTD. At the highest dose level 6 patients will be treated. The recommended dose for a phase II trial will be the lowest dose that results in the most effective VEGF neutralization, together with acceptable safety and toxicity.
  Interventions: Biological: hVEGF26-104/RFASE

INTERVENTIONS:
Biological: hVEGF26-104/RFASE — Three intramuscular injections on days 0, 14 and 28, followed by an observational period of 6 weeks. If hererafter VEGF is not (or no longer) neutralized in serum and there is no sign of disease progression, another booster vaccination can be given. This booster can be repeated until disease progression, death or withdrawal from the study.

SUMMARY:
The primary objectives of this study are to investigate the safety and tolerability profile of the therapeutic vaccine hVEGF26-104/RFASE and to determine the effective dose of hVEGF26-104/RFASE required to neutralize VEGF in serum, defined as a VEGF level below 9,0 pg/mL.

DETAILED DESCRIPTION:
Angiogenesis (the formation of new blood vessels from pre-existing blood vessels) plays an important role in the growth and spread of tumors. Angiogenesis is regulated by a balance of activators and inhibitors. One of the angiogenic activators is the vascular endothelial growth factor (VEGF, also referred to as VEGF-A). Over the past decade, several angiogenesis inhibitors have been discovered and implemented in the therapy of cancer patients. Bevacizumab (a humanized monoclonal antibody that inhibits VEGF-A) has been shown to improve survival in different tumor types in first and second line therapy when given in various chemotherapy combinations. Furthermore, research has shown a survival benefit of continued VEGF suppression with bevacizumab beyond first progression in metastatic colorectal cancer. So although repeated use of bevacizumab as a chronic therapy is much desired, currently this is not feasible because of substantial disadvantages of bevacizumab therapy. First, since bevacizumab only offers temporary VEGF neutralization, it needs frequent repeated administration. Secondly, bevacizumab is an intravenous therapy, which requires hospitalization on each administration. Third, bevacizumab has very high production costs. These specific drawbacks of longer term monoclonal antibody therapy could be circumvented by the use of a therapeutic cancer vaccine targeting VEGF. A vaccine is able to induce sustained VEGF suppression and can be administered via an intramuscular (IM) injection. In addition, a vaccine will likely inhibit VEGF more effectively as compared to bevacizumab, because a vaccine induces a polyclonal antibody response, resulting in higher avidity binding. Furthermore, it is believed that endogenous antibodies have a better tumor penetrating capacity, as compared to exogenously administered antibodies. The vaccine hVEGF26-104 is a truncated synthetic peptide mimic of the VEGF protein and consists of 79 amino acids (residue 26-104). The vaccine contains an antigen that directs the body's own polyclonal antibody response towards the active site of the endogenous VEGF molecule. After binding of the antibodies to endogenous VEGF this hormone will no longer be able to bind to its receptors (VEGFR1 and VEGFR2) and consequently will no longer exert its pro-angiogenic effect. To enhance the immune response, RFASE, which belongs to the adjuvant group of sulpholipopolysaccharides, will be used as an adjuvant.

Primary objectives - To investigate the safety and tolerability profile of hVEGF26-104/RFASE. - To determine the effective dose of hVEGF26-104/RFASE required to neutralize VEGF in serum, defined as a VEGF level below 9,0 pg/mL.

Secondary objectives - To determine the anti-VEGF antibody titer, induced by hVEGF26-104/RFASE administration. - To determine the effective dose of hVEGF26-104/RFASE required to neutralize VEGF in plasma and in a platelet sample. - To assess the effect of VEGF neutralization in a functional Ba/F3-R2 cell proliferation assay.

Exploratory objectives - To assess the cellular anti-tumor immune response induced by hVEGF26-104/RFASE administration. - To assess immunomodulatory effects upon hVEGF26-104/RFASE administration. - To make a preliminary assessment of hVEGF26-104/RFASE to suppress angiogenesis within the tumor. - To assess the immune infiltration and the regulation of endothelial cell adhesion molecules within the tumor.

This is an open label single center phase I study. A "3 + 3 " dose escalation design will be used. The study will investigate sequential cohorts consisting of 3 patients to be enrolled and treated at the applicable dose level. The study medication consists of 1.0 mL hVEGF26-104 (in escalating doses of 62.5, 125, 250 and 500 µg/mL) combined with 1.0 mL RFASE (fixed dose of 20 mg/mL). Eligible subjects will receive three IM injections with hVEGF26-104/RFASE on days 0 (primer), 14 and 28 (boosters). To assess potential toxicity of the adjuvant RFASE, the 3 patients enrolled in the first cohort of the study (62.5 μg/mL) will receive a single injection with 1.0 mL RFASE (fixed dose of 20 mg/mL) as a single agent 14 days prior to the first immunization with hVEGF26-104/RFASE. If none out of 3 patients experiences dose limiting toxicity (DLT) at a certain dose level, one can proceed to the next dose level. If one patient experiences a DLT at a certain dose level, another 3 patients will be assigned at the same dose level. In the highest dose escalation cohort, at least 6 patients will be enrolled. If VEGF is no longer neutralized, but there is no sign of progression either; the patient will receive another booster of hVEGF26-104/RFASE in order to achieve VEGF neutralization again. This booster can be repeated until progressive disease, death or other reasons for withdrawal from the study.

Eligible subjects will receive three intramuscular injections with hVEGF26-104/RFASE in dose-escalation on days 0 (primer), 14 and 28 (boosters), followed by an observation period of 6 weeks. Blood will be drawn at given timepoints to assess safety, immunogenicity and angiogenesis parameters. At screening, a tumor biopsy will be performed for a baseline assessment of angiogenesis and immune infiltration. In the case that VEGF is neutralized 8 weeks after first hVEGF26-104 administration, the patient will be asked to undergo another biopsy at week 10 to assess any possible change in angiogenesis and immune infiltration in the tumor. If VEGF is no longer neutralized, but there is no sign of progression either; the patient will receive another booster of hVEGF26-104/RFASE in order to achieve VEGF neutralization again.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced, solid malignancy.
* Refractory or not amenable to standard therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Please refer to Appendix II for more information.
* Willing and able to give written informed consent
* Patient is ≥ 18 years of age at the time of signature of the informed consent
* Adequate hematological function: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, Hemoglobin ≥ 6.0 mmol/L.
* Adequate hepatic function: serum bilirubin ≤ 1.5 times the upper limit of normal (ULN), ALT and AST ≤ 2.5 x ULN (or ≤ 5 times ULN if liver metastases are present).
* Adequate renal function: eGFR ≥ 50ml/min
* PT-INR/PTT < 1.5 x ULN, unless coumarin derivatives are used
* Activated partial thromboplastin time (APTT) < 1.25 x ULN (therapeutic anticoagulation therapy is allowed, if this treatment can be interrupted for a biopsy as judged by the treating physician)
* Female patients of childbearing potential may be enrolled in the study, if the patient

  * Has practiced adequate contraception for 30 days prior to first hVEGF26-104/RFASE administration.
  * Negative pregnancy test
  * Has agreed to continue adequate contraception for as long as VEGF is neutralized.

Exclusion Criteria:

* Major surgery within 28 days before the initiation of study treatment
* Any serious non-healing wounds, ulcers, or bone fractures within 28 days prior to the initiation of study treatment.
* Deep venous thrombosis (DVT) or pulmonary embolus (PE) within 1 year prior to the initiation of study treatment.
* Uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg)
* The patient is scheduled to receive another vaccination during the DLT period.
* A previous serious allergic reaction to a vaccine such as angioedema and anaphylaxis.
* Treatment with bevacizumab within 6 weeks prior to the initiation of study treatment.
* Uncontrolled auto-immune diseases
* Primary or secondary immunodeficiency, including HIV
* Treatment with a glucocorticoid derivative in an equivalent dose of ≥ 10mg prednisone a day.
* Female patients: the patient is pregnant or lactating.
* When the patient is scheduled to receive any other anticancer treatments.
* Chemotherapy within 28 days prior to the initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2020-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious and non-serious adverse events | 10-12 weeks
Neutralization of endogenous VEGF in serum | 10-12 weeks
  VEGF neutralization is defined as a VEGF level below 9,0 pg/mL as determined by sandwich ELISA.
Maximum tolerated dose (MTD) of hVEGF26-104/RFASE | 10-12 weeks

SECONDARY OUTCOMES:
Calculation of the anti-VEGF antibody titer in serum, plasma and a platelet sample | 10-12 weeks
Calculation of the functional VEGF neutralization. | 10-12 weeks
  Functional VEGF neutralization is defined as a significant decrease in cell proliferation as determined in a Ba/F3-R2 bioassay relative to pre-treatment values.
Neutralization of VEGF in plasma | 10-12 weeks
  VEGF neutralization is defined as a VEGF level below 9,0 pg/mL as determined by sandwich ELISA.

OTHER OUTCOMES:
Measurement of a cellular (T-cell) immune response, as determined by enzyme linked immunospot (ELISPOT) | 26 weeks
Measurement of immune modulation, through FACS analysis. | 26 weeks
Measuring angiogenesis suppression within the tumor. | 10-12 weeks
  This will be determined by assessing microvessel density (MVD), quantity of proliferating endothelial cells and pericyte coverage in tumor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Henk Verheul, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands